CLINICAL TRIAL: NCT06413407
Title: The Effect of Tai Chi Exercise and Receptive Music Therapy Applied to Elderly Individuals on Frailty Levels and Mental Health
Brief Title: Tai Chi Exercise and Receptive Music Therapy for the Elderly
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, NİHAN TÜRKOĞLU, Assist Prof., Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NihanT
Record Dates: First submitted 2024-05-09; First posted 2024-05-14 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Elderly; Exercise; Therapy
Keywords: Tai Chi Exercise; Receptive Music Therapy; Elderly; Vulnerability; Depression
MeSH Terms: conditions — Motor Activity; Depression | interventions — Aquatic Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Tai Chi Exercise Group (Active Comparator): As an intervention for this group, only Tai Chi Exercise will be applied.
  Interventions: Behavioral: Tai Chi Exercise
- Receptive Music Therapy Group (Active Comparator): As an intervention for this group, only Receptive Music Therapy Group will be applied.
  Interventions: Behavioral: Receptive Music Therapy
- Experimental (Experimental): As an intervention, both Tai Chi Exercise and Receptive Music Therapy will be applied to this group.
  Interventions: Behavioral: Experimental
- Control (No Intervention): No intervention will be applied to this group.

INTERVENTIONS:
Behavioral: Tai Chi Exercise — Tai Chi Exercise will be applied to this group.
  Arms: Tai Chi Exercise Group
Behavioral: Receptive Music Therapy — Receptive Music Therapy will be applied to this group.
  Arms: Receptive Music Therapy Group
Behavioral: Experimental — Tai Chi Exercise and Receptive Music Therapy techniques will be applied together to this group.
  Arms: Experimental

SUMMARY:
Frailty has become a major public health issue with the global aging population. In general, severe physical impairments and accompanying frailty in older adults are associated with adverse clinical outcomes. In addition to physical disorders, psychosocial disorders are also important in the formation of frailty. Depression is one of the most common psychosocial disorders among older adults, with prevalence ranging from 6.5% to 25.3%. Frail people may develop depression, and depressive symptoms negatively affect the physical functioning of the body, contributing to the development of frailty. This interrelationship between depression and frailty can lead to a vicious cycle with detrimental consequences for older adults. It is reported in the literature that elderly individuals experience low levels of well-being as well as depression. Spiritual well-being means that the individual is aware of his or her own abilities, feels at peace, is not affected by the stresses that may exist in his or her life, and is not in a state of spiritual turmoil. Poor mental health in the elderly increases fragility. This explains that frailty in elderly individuals affects all physical, social and psychological health components, and seriously negatively affects the quality of life and the formation and management of diseases. Most of the research literature on frailty has focused on physical health. But mental health, which includes positive aspects such as cognition, sleep, social interactions and well-being, is just as important as that related to physical illness and disability. There is a serious need for similar research focusing on psychosocial interventions to prevent and manage frailty. Studies are needed to show that promoting components such as resilience, social participation, and emotional regulation reduces stress levels in older adults, positively impacts mental health, increases healthy behaviors, and improves lifestyle, thereby reducing the risk of frailty. When the literature is evaluated, scientific studies in which music therapy and physical activity are applied have shown that these methods have positive effects on conditions that negatively affect mental health such as anxiety, stress and depression. There are no studies in the literature that discuss relaxing exercise and music therapy together for frailty in the elderly.

DETAILED DESCRIPTION:
The aim of this study is to determine the effect of relaxing exercise and music therapy on the level of fragility and mental health in the elderly, who are considered to be a risk group in terms of public health.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years or older
* Not having any obstacle to exercise
* He has no problems with his hearing

Exclusion Criteria:

* Not volunteering to participate in the study

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-15 (Estimated); Primary Completion 2024-08-15 (Estimated); Study Completion 2024-12-15 (Estimated)

PRIMARY OUTCOMES:
Depression, Anxiety, Stress Scale (DASS-21) | two week
  The four-point Likert-type scale developed by Lovibond and Lovibond (1995) consists of 14 depression, 14 anxiety and 14 stress dimensions; The short form of the scale, which consists of seven items each, consists of 21 items in order to have faster and more effective access to resources and more qualified use of time. It is presented in a four-point Likert form as "Not at All Appropriate (0) Somewhat Appropriate (1) Generally Appropriate (2) Completely Appropriate (4)" and shows that as the scores obtained from the scale increase, depression, anxiety and stress symptoms increase. Turkish validity and reliability studies were carried out by Yılmaz et al. Considering the reliability values, Cronbach's Alpha values for the dimensions are between 0.75-0.82; It is seen that the factor load Omega values for the dimensions are between 0.76 and 0.82 (Yılmaz et al., 2017).
Edmonton Frail Scale | Two week
  In order to evaluate frailty in the elderly, Rolfson et al. The validity and reliability study of the scale developed by Aygör in our country was carried out by Aygör. The scale consists of 11 questions and is evaluated in the range of 0-20 points. If the score obtained from the scale is in the range of 0-4, the elderly person is not fragile; A score of 5-6 is considered visibly vulnerable, a score of 7-8 is considered slightly fragile, a score of 9-10 is considered moderately fragile, and a score of 11 and above is considered severely fragile. In Aygör's study, the Cronbach alpha coefficient was determined as 0.75.

CONTACTS AND LOCATIONS:
Overall Officials: Nihan Türkoğlu, Principal Investigator — Ataturk University

IPD SHARING:
Plan to Share IPD: No